CLINICAL TRIAL: NCT06239519
Title: Increasing Access to Mental Health Support for 12-17 Year Old Youth With the JoyPop Mobile Mental Health App: Randomized Controlled Trial
Brief Title: JoyPop Mobile Mental Health App With Youth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lakehead University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 100157(2)
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Emotion Regulation; Depression; Anxiety; Stress
MeSH Terms: conditions — Emotional Regulation; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A pragmatic, parallel arm randomized controlled superiority trial will be used. Participants will be randomly allocated in a 1:1 ratio to the control (usual practice; UP) or intervention (UP + JoyPop) condition. Stratified block randomization (block size of 10) will be used to randomly assign participants to each condition.
Who Masked: Investigator
Masking Description: Given the nature of this trial, it will not be possible to blind participants to their allocation. As measures are self report, blinding of outcome measures is also not possible. Protect against bias will occur by blinding investigators to condition (i.e., only staff directly managing participants will be unblinded).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Practice + JoyPop (Experimental): Participants will be monitored through the existing wait-list practices, and will receive access to the JoyPop app for 4 weeks.
  Interventions: Behavioral: Usual Practice + JoyPop
- Usual Practice (No Intervention): Participants will be monitored through existing wait-list practices. After 4 weeks in the Usual Practice condition, participants will be offered access to the JoyPop app.

INTERVENTIONS:
Behavioral: Usual Practice + JoyPop — Participants will be asked to use the app at least twice daily but will otherwise not be provided with requirements related to feature or total usage.
  Arms: Usual Practice + JoyPop

SUMMARY:
Youth in Canada are in need of novel, innovative approaches to support their mental health and wellbeing. Within this age group, research suggests rates of several mental health difficulties and related hospitalizations have increased over recent decades. These challenges are exacerbated in rural communities, such as in Northwestern Ontario, where youth access mental health services less frequently and face longer wait times than those in more urban areas. Such limited access and extended waits can exacerbate symptoms, prolong distress, and increase the risk for adverse outcomes. In partnership with St. Joseph Care Group and Thunder Bay Counselling Centre, the investigators are evaluating the impact of a mental health app (JoyPop) as a tool for youth waiting for mental health services. The JoyPop app was developed to support improved emotion regulation - a fundamental difficulty for youth presenting with mental health challenges and an ability still undergoing maturation during this developmental period. A two-arm randomized controlled trial (RCT) will be used to evaluate the effectiveness of the app compared to usual practice while youth aged 12-17 are waiting for mental health services.

DETAILED DESCRIPTION:
Mental health services are less available and accessible in rural and northern communities than in urban areas. These issues are concerning as extended time on wait lists can exacerbate symptoms, prolong symptoms, prolong distress, and increase the risk for suicide, self-harm, and the need for hospitalization. Moreover, delayed access to mental health services negatively impacts treatment engagement, with non-attendance, decreased motivation, and reduced satisfaction with services frequently reported following prolonged wait times. A particularly vulnerable group in this context is adolescent youth, for whom research suggests mental health symptoms such as anxiety and depression and related hospital visits have increased in recent decades. Given the imminent need for and reduced access to accessible mental health services for youth in Northwestern Ontario, innovative solutions are needed. In partnership with St. Joseph Care Group and Thunder Bay Counselling Centre, the investigators are evaluating the impact of a mental health app (JoyPop) as a tool for youth who are waiting for mental health services. The JoyPop app was developed to support improved emotion regulation - an ability still undergoing development during adolescence and which can present as a key difficulty for youth with mental health challenges. Mobile mental health applications have the potential to increase accessible mental health support for youth in Northwestern Ontario. Despite this promise of mobile mental health apps, significant gaps exist between the growing number of apps available in the public domain and empirical evidence of the beneficial impacts of apps for users. In particular, most apps that focus on emotion regulation have not been evaluated, are narrow in scope, or have only been evaluated among adult populations. The JoyPop app includes a broader focus, and this research is unique given its focus on rigorously evaluating the JoyPop app as a tool for youth aged 12-17 in Northwestern Ontario, a population that has previously expressed interest in using the JoyPop in a pilot study.

Using a randomized controlled trial (RCT) design, the primary objective is to determine the effectiveness of the JoyPop app in improving emotion regulation among youth (12-17) who are waiting for mental health services as compared to usual practice (UP; monitoring those on the wait-list). The secondary objectives are to: (1) Assess change in mental health difficulties and treatment readiness between youth in each condition to better understand the app's broader impact as a wait-list tool; (2) Conduct an economic analysis to determine whether receiving the app while waiting for mental health services reduces other health service use and associated costs; (3) Define the Minimal Clinically Important Difference (MCID) for the primary outcome measure; and (4) Assess youth perspectives on the quality of the JoyPop app.

ELIGIBILITY:
Inclusion Criteria:

* Youth must be on the wait-list for mental health services at St. Joseph's Care Group or Thunder Bay Counselling Centre and be between 12-17 years old.
* Eligible youth will also need to be available to attend a virtual or in-person orientation session.
* In order to download the JoyPop app, participants will need access to an iOS device (e.g., iPhone, iPad). Refurbished iPhones containing just the JoyPop app will be provided to participants to use for the duration of the trial if they do not have access to their own.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in emotion regulation (overall) | Time Frame: Difficulties in Emotion Regulation Scale - Short Form will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Emotion regulation will be assessed with the Difficulties in Emotion Regulation Scale - Short Form. Total scores range from 18 to 90 with higher scores indicating greater difficulties in emotion regulation.
Change in emotion regulation (strategies) | Difficulties in Emotion Regulation Scale - Short Form will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Emotion regulation (strategies) will be assessed with the Difficulties in Emotion Regulation Scale - Short Form strategies subscale. Total scores range from 3 to 15 with higher scores indicating greater difficulties.
Change in emotion regulation (non-acceptance) | Difficulties in Emotion Regulation Scale - Short Form will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Emotion regulation (non-acceptance) will be assessed with the Difficulties in Emotion Regulation Scale - Short Form non-acceptance subscale. Total scores range from 3 to 15 with higher scores indicating greater difficulties.
Change in emotion regulation (impulse) | Difficulties in Emotion Regulation Scale - Short Form will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Emotion regulation (impulse) will be assessed with the Difficulties in Emotion Regulation Scale - Short Form impulse subscale. Total scores range from 3 to 15 with higher scores indicating greater difficulties.
Change in emotion regulation (goals) | Difficulties in Emotion Regulation Scale - Short Form will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Emotion regulation (goals) will be assessed with the Difficulties in Emotion Regulation Scale - Short Form goals subscale. Total scores range from 3 to 15 with higher scores indicating greater difficulties.
Change in emotion regulation (awareness) | Difficulties in Emotion Regulation Scale - Short Form will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Emotion regulation (awareness) will be assessed with the Difficulties in Emotion Regulation Scale - Short Form awareness subscale. Total scores range from 3 to 15 with higher scores indicating greater difficulties.
Change in emotion regulation (clarity) | Difficulties in Emotion Regulation Scale - Short Form will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Emotion regulation (clarity) will be assessed with the Difficulties in Emotion Regulation Scale - Short Form clarity subscale. Total scores range from 3 to 15 with higher scores indicating greater difficulties.

SECONDARY OUTCOMES:
Change in psychological distress | Depression Anxiety and Stress Scale 21 will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Psychological distress will be assessed with the total score for all items on the Depression Anxiety and Stress Scale 21. Total scores range from 0 to 63 with higher scores indicating greater psychological distress.
Change in depressive symptoms | Depression Anxiety and Stress Scale 21 will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Depressive symptoms will be assessed with the Depression subscale of the Depression Anxiety and Stress Scale 21. Total scores range from 0 to 21 with higher scores indicating greater depressive symptoms.
Change in anxious symptoms | Depression Anxiety and Stress Scale 21 will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Anxious symptoms will be assessed with the Anxiety subscale of the Depression Anxiety and Stress Scale 21. Total scores range from 0 to 21 with higher scores indicating greater anxious symptoms.
Change in stress | Depression Anxiety and Stress Scale 21 will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Stress will be assessed with the Stress subscale of the Depression Anxiety and Stress Scale 21. Total scores range from 0 to 21 with higher scores indicating greater stress symptoms.
Change in overall difficulties | Strengths and Difficulties Questionnaire will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Overall difficulties will be assessed with the total score from the Strengths and Difficulties Questionnaire (all subscales except prosocial). Total scores range from 0 to 40 with higher scores indicating worse difficulties.
Change in emotional problems | Strengths and Difficulties Questionnaire will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Emotional problems will be assessed with the Emotional Problems subscale from the Strengths and Difficulties Questionnaire. Total scores range from 0 to 10 with higher scores indicating worse emotional problems.
Change in conduct problems | Strengths and Difficulties Questionnaire will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Conduct problems will be assessed with the Conduct Problems subscale from the Strengths and Difficulties Questionnaire. Total scores range from 0 to 10 with higher scores indicating worse conduct problems.
Change in hyperactivity | Strengths and Difficulties Questionnaire will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Hyperactivity will be assessed with the Hyperactivity subscale from the Strengths and Difficulties Questionnaire. Total scores range from 0 to 10 with higher scores indicating worse hyperactivity.
Change in peer problems | Strengths and Difficulties Questionnaire will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Peer problems will be assessed with the Peer Problems subscale from the Strengths and Difficulties Questionnaire. Total scores range from 0 to 10 with higher scores indicating worse peer problems.
Change in prosocial behaviour | Strengths and Difficulties Questionnaire will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Prosocial behaviour will be assessed with the Prosocial subscale from the Strengths and Difficulties Questionnaire. Total scores range from 0 to 10 with lower scores indicating worse prosocial behaviour.
Change in treatment readiness | Treatment Readiness subscale of the Motivation for Youth's Treatment Scale will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Treatment readiness will be assessed with the Treatment Readiness subscale of the Motivation for Youth's Treatment Scale. Total scores range from 4 to 20 with higher scores indicating greater readiness.

OTHER OUTCOMES:
App quality (overall) | User Version of the Mobile Application Rating Scale will be administered to the intervention group after 4 weeks (post)
  App quality (overall) will be assessed with the User Version of the Mobile Application Rating Scale. Total scores range from 1 to 5 with higher scores indicating greater quality.
App quality (engagement) | User Version of the Mobile Application Rating Scale will be administered to the intervention group after 4 weeks (post)
  App quality (engagement) will be assessed with the Engagement subscale of the User Version of the Mobile Application Rating Scale. Total scores range from 1 to 5 with higher scores indicating greater quality (engagement).
App quality (functionality) | User Version of the Mobile Application Rating Scale will be administered to the intervention group after 4 weeks (post)
  App quality (functionality) will be assessed with the Functionality subscale of the User Version of the Mobile Application Rating Scale. Total scores range from 1 to 5 with higher scores indicating greater quality (functionality).
App quality (aesthetics) | User Version of the Mobile Application Rating Scale will be administered to the intervention group after 4 weeks (post)
  App quality (aesthetics) will be assessed with the Aesthetics subscale of the User Version of the Mobile Application Rating Scale. Total scores range from 1 to 5 with higher scores indicating greater quality (aesthetics).
App quality (information) | User Version of the Mobile Application Rating Scale will be administered to the intervention group after 4 weeks (post)
  App quality (information) will be assessed with the Information subscale of the User Version of the Mobile Application Rating Scale. Total scores range from 1 to 5 with higher scores indicating greater quality (information).
App quality (subjective) | User Version of the Mobile Application Rating Scale will be administered to the intervention group after 4 weeks (post)
  App quality (subjective) will be assessed with the Subjective subscale of the User Version of the Mobile Application Rating Scale. Total scores range from 1 to 5 with higher scores indicating greater quality (subjective).
App quality (perceived impact) | User Version of the Mobile Application Rating Scale will be administered to the intervention group after 4 weeks (post)
  App quality (perceived impact) will be assessed with the Perceived Impact subscale of the User Version of the Mobile Application Rating Scale. Total scores range from 1 to 5 with higher scores indicating greater quality (perceived impact).
Service utilization | Service utilization measure will be administered at baseline (pre), after 2 weeks (mid), and after 4 weeks (post)
  Service utilization will be assessed with 5 items asking about frequency of healthcare services accessed over the prior 2 weeks. Response options are open-ended and will be analyzed individually and as a total score across service types.
Minimal Clinically Important Difference (MCID) | GRC will be administered to the intervention group after 2 weeks (mid) and 4 weeks (post)
  On the Global Rating of Change (GRC), the smallest change in emotion regulation that participants identify as important after completing the trial will be used to calculate the MCID. The GRC is an 11-point Likert scale (ranging from -5 to +5; -5 very much worse, 0 unchanged, +5 very much better) used to indicate the degree to which emotion regulation changed for the better, for the worse, or no change after receiving the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Lakehead University, Thunder Bay, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No